



Title: Strength Training in Hypoxia to Improve Bone and Cardiovascular Health of Elderly

NCT number: not yet assigned

**Document Date: 25/May/2019** 





# **Brief Summary**

Due to age-related effects, the bone and cardiovascular health are damaged. Physical exercise and in particular the strength training has been proposed as a fundamental tool to these pathologies, especially in the elderly. On the other hand, the use of normobaric hypoxia combined with exercise could have a beneficial synergistic effect on disease prevention and the quality of life of the elderly.

Therefore, the general objective of this project is to analyze the effects of different methods of strength training combined with conditions of normobaric hypoxia on the bone and cardiovascular health of the elderly. This general objective is specified in the following specific objectives:

- To analyze the effects of resistance circuit training on bone mineral density and bone remodelling markers of elderly, under normoxic and normobaric hypoxic conditions.
- To analyze the effects of resistance circuit training on biochemical parameters, inflammatory, endothelial and clinical markers just like cardiovascular risk level of elderly, under normoxic and normobaric hypoxic conditions.
- To analyze the effects of resistance circuit training on body composition and functional capacity of elderly, under normoxic and normobaric hypoxic conditions.
- To analyze the effects of whole-body vibration training on bone mineral density and bone remodelling markers of elderly, under normoxic and normobaric hypoxic conditions.
- To analyze the effects of whole-body vibration training on biochemical parameters, inflammatory, endothelial and clinical markers just like cardiovascular risk level of elderly, under normoxic and normobaric hypoxic conditions.
- To analyze the effects of whole-body vibration training on body composition and functional capacity of elderly, under normoxic and normobaric hypoxic conditions.
- To compare the effects of resistance circuit versus whole-body vibration training on bone and cardiovascular health of elderly, under normoxic and normobaric hypoxic conditions.
- To value the normobaric hypoxic environment efficacy on bone and cardiovascular health of elderly subjected to resistance circuit and whole-body vibration training.

We hypothesize that bone and cardiovascular health will improve in the participants subjected to both resistance training, but greater improved may be found when these protocol are combined with normobaric hypoxia.





# Methodology

## **Participants**

Various associations of pensioners will be contacted as well as the university of seniors of the University of Extremadura to recruit volunteer participants. Total sample size will be 120 people, being this calculated to obtaining a statistical power of 90%, calculated with a margin of error of 5% and a mean difference of 10% in the study variables.

Inclusion criteria will be: (1) women and men aged 65 years or older; (2) no current medical condition not compatible with planned exercise; (3) free of illness or medication potentially affecting the bone and cardiovascular system; (4) estimated daily calcium intake of 1200-2000 mg/day; (5) consumption of no more than two alcoholic beverages per day. Exclusion criteria will be: (1) participation in any other type of intervention based on physical exercise in the last 6 months in order to avoid interactions with the previous practice; (2) subjects have been above 1500 m during the last 3 months; (3) contra indications for whole-body vibration training: severe cardiovascular diseases, ocular diseases that affect the retina, neuromuscular and heart diseases, stroke, implant, bypass, stent, arthritis and other joint disease or epilepsy.

Participants will be assigned to 6 different groups: (1) Normoxia Control Group (NCON), who will be instructed to continue with their normal daily activities for the entire duration of the study; (2) Hypoxia Control Group (HCON); who will perform an intellectual activity while they will be exposed to normobaric hypoxic conditions (16.0% FiO2); (3) Normoxia Circuit Training (NCIR); who will perform a circuit training with elastic bands in normoxic conditions (20.9% FiO2); (4) Hypoxia Circuit Training (HCIR); who will perform a circuit training with elastic bands in hypoxic conditions (16.0% FiO2); (5) Normoxia Vibration (NVIB); who will perform whole-body vibration training in normoxic conditions (20.9% FiO2); (6) Hypoxia Vibration (HVIB); who will perform whole-body vibration training in hypoxic conditions (16.0% FiO2).

All procedures will be performed in studies involving human participants will be in accordance with the 1964 Helsinki declaration and its later amendments or comparable ethical standards and the study design was approved by the Bioethical and Biosecurity Commission of the University of Extremadura (65/2018).

#### Design

This will be a randomised double-blind controlled study. There were separate intervention and assessment teams. We will try to blind the study for participants, as they will be trained/tested separately. Training sessions will be supervised by an experienced member of the research group.

All interventions will be performed during 24 weeks, with a frequency training of 3 days per weeks; sessions will be scheduled with at least one day of rest in between for optimal recovery. All patients were assessed at two time points: at baseline before the 24 weeks of intervention (Pre) and reassessed 7 days after the last session (Post). Participants will be instructed to continue with their normal daily activities, diet and caloric and calicium intake for the entire duration of the study.

#### Interventions

During several times of the session in each intervention, oxygen saturation (SpO<sub>2</sub>) will be controlled using a finger pulse-oximeter (Konica Minolta, Japan) and heart rate (HR)





using a heart rate monitor (Polar team 2, Polar, Finland) to know the physiological challenge posed on the participants during the exposure.

#### Passive hypoxia

During 30 minutes of session, the participants will be performed an intellectual activity while they will be exposed to normobaric hypoxic conditions in a hypoxic chamber (CAT 310, Lousiville, Colorado). They will inspire oxygen fraction (FiO2) set to 16.1% (0.16) in order to simulate an altitude of 2500m above sea level.

#### Normoxia circuit training

Each training sessions will consist of a circuit training with elastic bands, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit that will be composed by 3 sets of 12-15 repetitions of nine different exercises. Six exercises will be performed using elastic resistance bands (ERS; TheraBand®): chest press, row, glute kickbacks, front and side raises, standing biceps curls and triceps kickbacks. To provide resistance with ERB, elastic bands with resistance ranging from light to very heavy loading (colors: vellow-gold) were used. ERBs were 2 meters, but the actual length used (grip on ERBs and distance to anchor point) was fine tuned for each subject in each exercise to find the correct resistance. When necessary to increase loading, two or more bands were combined. Bands were prestretched and never elongated more than 300% of resting length, as recommended by the manufacturer. Two additional exercise will be developed with kettlebell (KB): squat with 6 kg or increase loading until 10 kg; and hip trust, increase loading with support of a foot alone or with additional loading (KB of 5 or 10 kg). Finally, the subjects will keep a plank position during 15-20 seconds.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. In order to blind subjects to altitude, the system will be run with normoxic airflow into the chamber (up to 1000 l/min) and will produce the same audible noise as in the hypoxic condition. Subjects will inspire FiO2 of 21.0% (0.21) to simulate an altitude of 459 m above sea level. Furthermore, all systems will be covered with fabric to prevent participants from visually identifying the normoxic or hypoxic conditions. FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).

## Hypoxia circuit training

Each training sessions will consist of a circuit training with elastic bands, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit, that will be composed by 3 sets of 12-15 repetitions of nine different exercises. Six exercises will be performed using elastic resistance bands (ERS; TheraBand®): chest press, row, glute kickbacks, front and side raises, standing biceps curls and triceps kickbacks. To provide resistance with ERB, elastic bands with resistance ranging from light to very heavy loading (colors: yellow-gold) were used. ERBs were 2 meters, but





the actual length used (grip on ERBs and distance to anchor point) was fine tuned for each subject in each exercise to find the correct resistance. When necessary to increase loading, two or more bands were combined. Bands were prestretched and never elongated more than 300% of resting length, as recommended by the manufacturer. Two additional exercise will be developed with kettlebell (KB): squat with 6 kg or increase loading until 10 kg; and hip trust, increase loading with support of a foot alone or with additional loading (KB of 5 or 10 kg). Finally, the subjects will keep a plank position during 15-20 seconds

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. Participants will inspire a fraction of inspired oxygen (FiO2) of 16.1% (0.16) to simulate an altitude of 2500 m above sea level; FiO2 will be controlled regularly with an electronic device (HANDIC, Maxtec, Salt Lake City, Utah, United States).

### Normoxia whole-body vibration

The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the session.

Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1–12 and 45 seconds between 5 repetitions during weeks 12–24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performance, with the soles of both feet remained in contact with the platform:

- 1) Stand with feet side-by-side on the board, which produced lateral oscillations of the whole body. During the vibration training sessions, the subjects will be barefoot to eliminate any damping of the vibration caused by footwear. The angle of flexion of the knees during the vibration exercise will be set at 60°.
- 2) Begin with the feet placed perpendicular to the midline axis of the platform, with a foot positioned slightly ahead of the other foot. Lift the toes of the one foot and the heel of the other foot 4 mm above the surface of the platform. Bend the knees and maintain a 45°knee angle. Keep the back and head straight. Alternate legs.
- 3) Front foot 4 mm above the surface of the platform and back foot on ground, front knee angle 90°. Alternate legs
- 4) Lay down on the ground, with the knees bent and feet flat on the platform. Keep the arms at your side with your palms down. Lift the hips off the ground until the knees, hips and shoulders form a straight line. Hold your bridged position.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. In order to blind subjects to altitude, the system will be run with normoxic airflow into the chamber (up to 1000 l/min) and will produce the same audible noise as in the hypoxic condition. Subjects will inspire FiO2 of 21.0% (0.21) to simulate an altitude of 459 m above sea level. Furthermore, all systems will be covered with fabric to prevent participants from visually identifying the normoxic or hypoxic conditions. FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).





## Hypoxia whole-body vibration

The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the session.

Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1–12 and 45 seconds between 5 repetitions during weeks 12–24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performance, with the soles of both feet remained in contact with the platform:

- 1) Stand with feet side-by-side on the board, which produced lateral oscillations of the whole body. During the vibration training sessions, the subjects will be barefoot to eliminate any damping of the vibration caused by footwear. The angle of flexion of the knees during the vibration exercise will be set at 60°.
- 2) Begin with the feet placed perpendicular to the midline axis of the platform, with a foot positioned slightly ahead of the other foot. Lift the toes of the one-foot and the heel of the other foot 4 mm above the surface of the platform. Bend the knees and maintain a 45°knee angle. Keep the back and head straight. Alternate legs.
- 3) Front foot 4 mm above the surface of the platform and back foot on ground, front knee angle 90°. Alternate legs
- 4) Lay down on the ground, with the knees bent and feet flat on the platform. Keep the arms at your side with your palms down. Lift the hips off the ground until the knees, hips and shoulders form a straight line. Hold your bridged position.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. Participants will inspire a fraction of inspired oxygen (FiO2) of 16.1% (0.16) to simulate an altitude of 2500 m above sea level; FiO2 will be controlled regularly with an electronic device (HANDIC, Maxtec, Salt Lake City, Utah, United States).

#### **Outcome Measures**

Socio-Demographic Data and Lifestyle Questionnaires

A general questionnaire was administered to collect medical and demographic data to check the inclusion/exclusion criteria. As control variables, prior and after the intervention, calcium intake was estimated using a food frequency questionnaire. The bone-specific physical activity questionnaire (B-PAQ) was used to assess the physical activity level of the participants in the last 12 months.

### Life Quality and Risk of Fall Questionnaires

SF-36 questionnaire will be used to know the life quality. Risk of fall will be evaluated through Fall Efficacy Scale-International (FES-I).

#### Cardiovascular Evaluation

Clinical tests of cardiovascular evaluation, such as recording of blood pressure with sphygmomanometer, arm-ankle index and pulse wave velocity using ultrasound Doppler technique will be used.





#### Cardiovascular Risk

Cardiovascular risk will be determined based on the following factors: age, sex, smoking, total cholesterol, HDL cholesterol, systolic blood pressure and diabetes, as described in the FRESCO study.

### Anthropometric Measurements

Weight, height, body mass index and waist-hip ratio will measure following standart procedures.

#### Body composition

Body composition variables such as percentage fat, lean and bone mass will be obtain using dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States) of whole body and corporal segment.

### Bone Mineral Density

Bone mineral content (g) and density (g/cm-2) and T-score of whole body and proximal femur region will be calculated from obtained data of dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States)

#### **Blood Biomarkers**

Standard biochemical analysis (HDL, LDL and Total Cholesterol, Triglycerides and Glucose) will be obtained of blood samples, through a clinical chemistry analyzer (Spotchem, Arkray Factory, Germany). Bone remodelling (VEGF and SDF-1), inflammatory (C-reactive protein, IL-2, IL-4, IL-6 and TNF alfa) and endothelial (ICAM-1 and VCAM-1) markers will be analyzed by ELISA technique.

### Functional Capacity

Senior Fitness Test battery will be used to know of physical condition of elderly: lower limb strength (Chair stand), upper limb strength (Arm curl), lower limb flexibility (Chair sit and reach), upper limb flexibility (Back scratch), endurance (6 min. walk) and agility (8ft Up and Go) will be tested through this battery. Furthermore, core muscle strength (plank test), grip strength (hand grip) and balance (single leg stance test) will be measured





# **Statistical Analysis Plan (SAP)**

Statistical analyses will be performed using the statistical analysis package SPSS v.20 (IBM, New York, United States). Data will be expressed as median and standard deviation. Kolmogorov–Smirnov tests will be conducted to show the distribution of the studied variables and Levene's test for homogeneity of variance. Repeated measure ANOVA will be used to compare the response of each variable, considering the sex and age as covariate. The p < 0.05 criterion was used for establishing statistical significance. Effect size (Cohen, 1992) will be also calculated for all variables, considering the magnitude of change as small (0.2), moderate (0.5) or large (0.8).





## References

- Bhella, P. S., Hastings, J. L., Fujimoto, N., Shibata, S., Carrick-Ranson, G., Palmer, M. D., . . . Levine, B. D. (2014). Impact of lifelong exercise "dose" on left ventricular compliance and distensibility. *J Am Coll Cardiol*, 64(12), 1257-1266. doi: 10.1016/j.jacc.2014.03.062
- Bliuc, D., Nguyen, N. D., Milch, V. E., Nguyen, T. V., Eisman, J. A., & Center, J. R. (2009). Mortality risk associated with low-trauma osteoporotic fracture and subsequent fracture in men and women. *JAMA*, 301(5), 513-521. doi: 10.1001/jama.2009.50
- Bogaerts, A., Delecluse, C., Boonen, S., Claessens, A. L., Milisen, K., & Verschueren, S. M. (2011). Changes in balance, functional performance and fall risk following whole body vibration training and vitamin D supplementation in institutionalized elderly women. A 6 month randomized controlled trial. *Gait Posture*, 33(3), 466-472. doi: 10.1016/j.gaitpost.2010.12.027
- Buckinx, F., Beaudart, C., Maquet, D., Demonceau, M., Crielaard, J. M., Reginster, J. Y., & Bruyere, O. (2014). Evaluation of the impact of 6-month training by whole body vibration on the risk of falls among nursing home residents, observed over a 12-month period: a single blind, randomized controlled trial. *Aging Clin Exp Res*, 26(4), 369-376. doi: 10.1007/s40520-014-0197-z
- Burghardt, A. J., Buie, H. R., Laib, A., Majumdar, S., & Boyd, S. K. (2010). Reproducibility of direct quantitative measures of cortical bone microarchitecture of the distal radius and tibia by HR-pQCT. *Bone*, 47(3), 519-528. doi: 10.1016/j.bone.2010.05.034
- Celis-Morales, C. A., Welsh, P., Lyall, D. M., Steell, L., Petermann, F., Anderson, J., . . . Gray, S. R. (2018). Associations of grip strength with cardiovascular, respiratory, and cancer outcomes and all cause mortality: prospective cohort study of half a million UK Biobank participants. *BMJ*, 361, k1651. doi: 10.1136/bmj.k1651
- Cenzer, I. S., Tang, V., Boscardin, W. J., Smith, A. K., Ritchie, C., Wallhagen, M. I., . . . Covinsky, K. E. (2016). One-Year Mortality After Hip Fracture: Development and Validation of a Prognostic Index. *J Am Geriatr Soc*, 64(9), 1863-1868. doi: 10.1111/jgs.14237
- Chan, D. A., Sutphin, P. D., Denko, N. C., & Giaccia, A. J. (2002). Role of prolyl hydroxylation in oncogenically stabilized hypoxia-inducible factor-1alpha. *J Biol Chem*, 277(42), 40112-40117. doi: 10.1074/jbc.M206922200
- Cummings, S. R., & Melton, L. J. (2002). Epidemiology and outcomes of osteoporotic fractures. *Lancet*, *359*(9319), 1761-1767. doi: 10.1016/S0140-6736(02)08657-9
- Delecluse, C., Roelants, M., & Verschueren, S. (2003). Strength increase after whole-body vibration compared with resistance training. *Med Sci Sports Exerc*, 35(6), 1033-1041. doi: 10.1249/01.MSS.0000069752.96438.B0
- Dreimuller, N., Schlicht, K. F., Wagner, S., Peetz, D., Borysenko, L., Hiemke, C., . . . Tadic, A. (2012). Early reactions of brain-derived neurotrophic factor in plasma (pBDNF) and outcome to acute antidepressant treatment in patients with Major Depression. *Neuropharmacology*, 62(1), 264-269. doi: 10.1016/j.neuropharm.2011.07.017
- Erickson, K. I., Voss, M. W., Prakash, R. S., Basak, C., Szabo, A., Chaddock, L., . . . Kramer, A. F. (2011). Exercise training increases size of hippocampus and improves memory. *Proc Natl Acad Sci U S A*, 108(7), 3017-3022. doi: 10.1073/pnas.1015950108
- Fratini, A., Bonci, T., & Bull, A. M. (2016). Whole Body Vibration Treatments in Postmenopausal Women Can Improve Bone Mineral Density: Results of a Stimulus Focussed Meta-Analysis. *PLoS One*, 11(12), e0166774. doi: 10.1371/journal.pone.0166774
- Gianoudis, J., Bailey, C. A., Ebeling, P. R., Nowson, C. A., Sanders, K. M., Hill, K., & Daly, R. M. (2014). Effects of a targeted multimodal exercise program incorporating high-speed power training on falls and fracture risk factors in older adults: a community-based randomized controlled trial. *J Bone Miner Res*, 29(1), 182-191. doi: 10.1002/jbmr.2014
- Gonzalez-Aguero, A., Vicente-Rodriguez, G., Gomez-Cabello, A., & Casajus, J. A. (2013). Cortical and trabecular bone at the radius and tibia in male and female adolescents with Down syndrome: a peripheral quantitative computed tomography (pQCT) study. *Osteoporos Int, 24*(3), 1035-1044. doi: 10.1007/s00198-012-2041-7





- Goudarzian, M., Ghavi, S., Shariat, A., Shirvani, H., & Rahimi, M. (2017). Effects of whole body vibration training and mental training on mobility, neuromuscular performance, and muscle strength in older men. *J Exerc Rehabil*, *13*(5), 573-580. doi: 10.12965/jer.1735024.512
- Goudarzian, M., Rahimi, M., Karimi, N., Samadi, A., Ajudani, R., Sahaf, R., & Ghavi, S. (2017). Mobility, Balance, and Muscle Strength Adaptations to Short-Term Whole Body Vibration Training Plus Oral Creatine Supplementation in Elderly Women. *Asian J Sports Med*, 8(1), e36793. doi: 10.5812/asjsm.36793.
- Graham, I., Atar, D., Borch-Johnsen, K., Boysen, G., Burell, G., Cifkova, R., . . . European Atherosclerosis, Society. (2007). European guidelines on cardiovascular disease prevention in clinical practice: full text. Fourth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts). *Eur J Cardiovasc Prev Rehabil*, 14 Suppl 2, S1-113. doi: 10.1097/01.hjr.0000277983.23934.c9
- Guner, Ibrahim, Uzun, Duygu D., Yaman, Muhittin O., Genc, Habibe, Gelisgen, Remisa, Korkmaz, Gulcan G., . . . Simsek, Gonul. (2013). The effect of chronic long-term intermittent hypobaric hypoxia on bone mineral density in rats: role of nitric oxide. *Biol Trace Elem Res, 154*(2), 262-267.
- Hinton, P. S., Nigh, P., & Thyfault, J. (2015). Effectiveness of resistance training or jumping-exercise to increase bone mineral density in men with low bone mass: A 12-month randomized, clinical trial. *Bone*, 79, 203-212. doi: 10.1016/j.bone.2015.06.008
- Inness, M. W., Billaut, F., Walker, E. J., Petersen, A. C., Sweeting, A. J., & Aughey, R. J. (2016). Heavy Resistance Training in Hypoxia Enhances 1RM Squat Performance. *Front Physiol*, 7, 502. doi: 10.3389/fphys.2016.00502
- Johnell, O., & Kanis, J. (2005). Epidemiology of osteoporotic fractures. *Osteoporos Int, 16 Suppl 2*, S3-7. doi: 10.1007/s00198-004-1702-6
- Johnell, O., & Kanis, J. A. (2006). An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int, 17(12), 1726-1733. doi: 10.1007/s00198-006-0172-4
- Kawanabe, K., Kawashima, A., Sashimoto, I., Takeda, T., Sato, Y., & Iwamoto, J. (2007). Effect of whole-body vibration exercise and muscle strengthening, balance, and walking exercises on walking ability in the elderly. *Keio J Med*, *56*(1), 28-33.
- Kon, M., Ohiwa, N., Honda, A., Matsubayashi, T., Ikeda, T., Akimoto, T., . . . Russell, A. P. (2014). Effects of systemic hypoxia on human muscular adaptations to resistance exercise training. *Physiol Rep*, 2(6). doi: 10.14814/phy2.12033
- Kraemer, W. J., Ratamess, N. A., & French, D. N. (2002). Resistance training for health and performance. *Curr Sports Med Rep, 1*(3), 165-171.
- McMillan, L. B., Zengin, A., Ebeling, P. R., & Scott, D. (2017). Prescribing Physical Activity for the Prevention and Treatment of Osteoporosis in Older Adults. *Healthcare (Basel)*, 5(4). doi: 10.3390/healthcare5040085
- Mikhael, M., Orr, R., Amsen, F., Greene, D., & Singh, M. A. (2010). Effect of standing posture during whole body vibration training on muscle morphology and function in older adults: a randomised controlled trial. *BMC Geriatr*, 10, 74. doi: 10.1186/1471-2318-10-74
- Navarrete-Opazo, A., & Mitchell, G. S. (2014). Therapeutic potential of intermittent hypoxia: a matter of dose. *Am J Physiol Regul Integr Comp Physiol*, 307(10), R1181-1197. doi: 10.1152/ajpregu.00208.2014
- Niino, N., Tsuzuku, S., Ando, F., & Shimokata, H. (2000). Frequencies and circumstances of falls in the National Institute for Longevity Sciences, Longitudinal Study of Aging (NILS-LSA). *J Epidemiol, 10*(1 Suppl), S90-94.
- Papa, E. V., Foreman, K. B., & Dibble, L. E. (2015). Effects of age and acute muscle fatigue on reactive postural control in healthy adults. *Clin Biomech (Bristol, Avon)*, 30(10), 1108-1113. doi: 10.1016/j.clinbiomech.2015.08.017





- Papa, E. V., Garg, H., & Dibble, L. E. (2015). Acute effects of muscle fatigue on anticipatory and reactive postural control in older individuals: a systematic review of the evidence. *J Geriatr Phys Ther*, 38(1), 40-48. doi: 10.1519/JPT.000000000000000006
- Pouyssegur, J., Dayan, F., & Mazure, N. M. (2006). Hypoxia signalling in cancer and approaches to enforce tumour regression. *Nature*, 441(7092), 437-443. doi: 10.1038/nature04871
- Rubin, C., Recker, R., Cullen, D., Ryaby, J., McCabe, J., & McLeod, K. (2004). Prevention of postmenopausal bone loss by a low-magnitude, high-frequency mechanical stimuli: a clinical trial assessing compliance, efficacy, and safety. *J Bone Miner Res*, 19(3), 343-351. doi: 10.1359/JBMR.0301251
- Rubin, C., Turner, A. S., Mallinckrodt, C., Jerome, C., McLeod, K., & Bain, S. (2002). Mechanical strain, induced noninvasively in the high-frequency domain, is anabolic to cancellous bone, but not cortical bone. *Bone*, 30(3), 445-452.
- Sallis, R. (2015). Exercise is medicine: a call to action for physicians to assess and prescribe exercise. *Phys Sportsmed*, 43(1), 22-26. doi: 10.1080/00913847.2015.1001938
- Schega, L., Peter, B., Torpel, A., Mutschler, H., Isermann, B., & Hamacher, D. (2013). Effects of intermittent hypoxia on cognitive performance and quality of life in elderly adults: a pilot study. *Gerontology*, 59(4), 316-323. doi: 10.1159/000350927
- Scott, B. R., Slattery, K. M., Sculley, D. V., & Dascombe, B. J. (2014). Hypoxia and resistance exercise: a comparison of localized and systemic methods. *Sports Med*, 44(8), 1037-1054. doi: 10.1007/s40279-014-0177-7
- Shaw, B. S., Shaw, I., & Mamen, A. (2010). Contrasting effects in anthropometric measures of total fatness and abdominal fat mass following endurance and concurrent endurance and resistance training. *J Sports Med Phys Fitness*, 50(2), 207-213.
- Shaw, I., Shaw, B. S., Brown, G. A., & Cilliers, J. F. (2010). Concurrent resistance and aerobic training as protection against heart disease. *Cardiovasc J Afr.*, 21(4), 196-199.
- Sipila, S., Elorinne, M., Alen, M., Suominen, H., & Kovanen, V. (1997). Effects of strength and endurance training on muscle fibre characteristics in elderly women. *Clin Physiol*, 17(5), 459-474
- Swanson, C. M., Shea, S. A., Stone, K. L., Cauley, J. A., Rosen, C. J., Redline, S., . . . Orwoll, E. S. (2015). Obstructive sleep apnea and metabolic bone disease: insights into the relationship between bone and sleep. *J Bone Miner Res*, 30(2), 199-211. doi: 10.1002/jbmr.2446
- Tosteson, A. N., Gottlieb, D. J., Radley, D. C., Fisher, E. S., & Melton, L. J., 3rd. (2007). Excess mortality following hip fracture: the role of underlying health status. *Osteoporos Int, 18*(11), 1463-1472. doi: 10.1007/s00198-007-0429-6
- von Friesendorff, M., McGuigan, F. E., Wizert, A., Rogmark, C., Holmberg, A. H., Woolf, A. D., & Akesson, K. (2016). Hip fracture, mortality risk, and cause of death over two decades. *Osteoporos Int*, 27(10), 2945-2953. doi: 10.1007/s00198-016-3616-5
- Watson, S. L., Weeks, B. K., Weis, L. J., Horan, S. A., & Beck, B. R. (2015). Heavy resistance training is safe and improves bone, function, and stature in postmenopausal women with low to very low bone mass: novel early findings from the LIFTMOR trial. *Osteoporos Int, 26*(12), 2889-2894. doi: 10.1007/s00198-015-3263-2
- Westcott, W. L. (2012). Resistance training is medicine: effects of strength training on health. *Curr Sports Med Rep*, 11(4), 209-216. doi: 10.1249/JSR.0b013e31825dabb8
- Williams, A. D., Almond, J., Ahuja, K. D., Beard, D. C., Robertson, I. K., & Ball, M. J. (2011). Cardiovascular and metabolic effects of community based resistance training in an older population. *J Sci Med Sport*, 14(4), 331-337. doi: 10.1016/j.jsams.2011.02.011
- Winklmayr, M., Kluge, C., Winklmayr, W., Kuchenhoff, H., Steiner, M., Ritter, M., & Hartl, A. (2015). Radon balneotherapy and physical activity for osteoporosis prevention: a randomized, placebocontrolled intervention study. *Radiat Environ Biophys*, *54*(1), 123-136. doi: 10.1007/s00411-014-0568-z
- Yang, Y. Q., Tan, Y. Y., Wong, R., Wenden, A., Zhang, L. K., & Rabie, A. B. (2012). The role of vascular endothelial growth factor in ossification. *Int J Oral Sci*, 4(2), 64-68. doi: 10.1038/ijos.2012.33





- Zaki, M. E. (2014). Effects of whole body vibration and resistance training on bone mineral density and anthropometry in obese postmenopausal women. *J Osteoporos*, 2014, 702589. doi: 10.1155/2014/702589
- Zhang, L., Weng, C., Liu, M., Wang, Q., Liu, L., & He, Y. (2014). Effect of whole-body vibration exercise on mobility, balance ability and general health status in frail elderly patients: a pilot randomized controlled trial. *Clin Rehabil*, 28(1), 59-68. doi: 10.1177/0269215513492162
- Zhao, R., Zhao, M., & Xu, Z. (2015). The effects of differing resistance training modes on the preservation of bone mineral density in postmenopausal women: a meta-analysis. *Osteoporos Int*, 26(5), 1605-1618. doi: 10.1007/s00198-015-3034-0
- Zuo, C., Huang, Y., Bajis, R., Sahih, M., Li, Y. P., Dai, K., & Zhang, X. (2012). Osteoblastogenesis regulation signals in bone remodeling. *Osteoporos Int*, 23(6), 1653-1663. doi: 10.1007/s00198-012-1909-x